CLINICAL TRIAL: NCT05944900
Title: Randomized, Prospective, Single-center Trial Comparing the Efficacy of Peripherally Inserted Central Catheter (PICC) Placement With the Addition of Cyanoacrylate Glue Versus PICC Placement Alone (Without Glue) in Patients With Cancer.
Brief Title: Study Comparing the Efficacy of Peripherally Inserted Central Catheter (PICC) Placement With the Addition of Cyanoacrylate Glue Versus PICC Placement Alone in Patients With Cancer.
Acronym: PICCandGLUE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Leon Berard (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: ET23-122
Record Dates: First submitted 2023-07-05; First posted 2023-07-13 (Actual); Last update posted 2024-09-27 (Actual); Status verified 2024-09

CONDITIONS: Cancer
Keywords: Cancer; Peripherally Inserted Central Catheter (PICC); Cyanoacrylate Glue
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Intervention Model Description: The randomization (1:1 ratio) will be stratified according to the risk of haemostasis disorders (Presence of at least one risk factor (medication interfering with hemostasis, innate or acquired coagulation disorder, thrombocytopenia) vs. no risk).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PICC placement according to standard practice + cyanoacrylate glue (Experimental): PICC placement will be performed according to standard practice (Safe Insertion of PICC protocol (SIP2) steps).
  The catheter will be secured by the Statlock system. Cyanoacrylate glue will be applied on the catheter exit point in accordance with the instructions for use.
  A transparent dressing will be applied, with a compress in the event of bleeding.
  Interventions: Procedure: Cyanoacrylate glue application
- PICC placement according to standard practice (No Intervention): PICC placement will be performed according to standard practice (Safe Insertion of PICC protocol (SIP2) steps).
  The catheter will be secured by the Statlock system. A transparent dressing will be applied, with a compress in the event of bleeding.

INTERVENTIONS:
Procedure: Cyanoacrylate glue application — The wound must be positioned in a horizontal plane, and the glueapplied uniformly overhanging the wound. Cyanoacrylate glue is contraindicated when adhesion cannot be achieved.
  Cyanoacrylate glue should be applied in accordance with the instructions for use.
  Wound-closing properties are only fully achieved once the first layer has fully polymerized. This depends on skin type, skin hydration and ambient humidity. If a second layer is applied, the polymerization time is extended accordingly.
  Arms: PICC placement according to standard practice + cyanoacrylate glue

SUMMARY:
This is a randomized, prospective, single-center trial comparing the efficacy of peripherally inserted central catheter (PICC) with the addition of cyanoacrylate glue versus PICC placement alone (without glue) in cancer patients.

DETAILED DESCRIPTION:
Peripherally Inserted Central Catheters (PICCs) are a form of vascular access inserted percutaneously into a vein, usually in the arm, with the distal end at the atrio cava junction (between the superior vena cava and the right atrium). They may be used for a prolonged period or for several days, repeatedly over time (as is the case for certain chemotherapies, parenteral nutrition or long-term intravenous treatments).

Their placement requires aseptic surgical conditions, and a team trained in the procedure, sometimes grouped together in a Vascular Access Unit (UAV).

A PICC is inserted by puncturing the skin and subcutaneous tissues, and securing the catheter with a "Statlock" type stabilizer. The catheter exit point must be covered, at a minimum by a sterile occlusive dressing with a transparent semi-permeable membrane, otherwise referred to as a "transparent dressing".

According to available data, tissue puncture results in bleeding at the puncture site in 25% to 40% of procedures. This bleeding necessitates the application of a sterile compress prior to covering with a transparent dressing. The skin puncture site (also known as the catheter exit point) requires the dressing to be repeated on D1 after insertion.

To sum up:

* If there is no bleeding, there is no need to apply a compress, and the dressing can be changed on D8 after application;
* In the presence of bleeding, a compress is applied and dressing change is mandatory on D1 after application.

PICC placement combined with the use of cyanoacrylate glue would reduce the risk of bleeding, and therefore the need to use of a compress, compared with a standard procedure (without the use of glue).

On this basis, the investigators propose to conduct a randomized, prospective, single-center trial comparing the efficacy of peripherally inserted central catheter (PICC) with the addition of cyanoacrylate glue versus PICC placement alone (without glue) in patients with cancer.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, 18 years of age or older on the date of signature the informed consent form
* Patient with a histological diagnosis of cancer
* Indication for central line chemotherapy or immunotherapy
* Placement of a single-lumen PICC in the non-tunneled upper limb planned on an ambulatory basis at the Centre
* Planned duration of PICC use > 30 days
* Dated and signed informed consent, indicating that the patient has been informed of all relevant aspects of the study prior to inclusion;
* Patient covered by a health insurance plan

Exclusion Criteria:

* Patient already included in the study ;
* Patient with known allergy to cyanoacrylates, Violet D&C or formaldehyde;
* Patient not reachable by telephone ;
* Patient under guardianship;
* Patient does not speak French.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2023-08-02 (Actual); Primary Completion 2024-06-19 (Actual); Study Completion 2024-07-19 (Actual)

PRIMARY OUTCOMES:
Rate of patients with successful PICC placement | Hour 0
  Success is defined by the possibility of using a dressing without compression at application (at hour 0), i.e. without bleeding after the defined compression time.

SECONDARY OUTCOMES:
Proportion of dressing changes within one hour | Up to hour 1
  Proportion of patients requiring dressing changes at the CLB within one hour of the end of procedure
Proportion of dressing changes before day 8 | Up to day 8
  Proportion of patients requiring dressing changes (home nursing/home care/home hospitalization) in the medium term (day 8)
Proportion of dressing changes before day 30 | Up to day 30
  Proportion of patients requiring dressing changes (home nursing/home care/home hospitalization) in the medium term (day 30)
Incidence of PICC removal before day 30 | Up to day 30
  Incidence of PICC removal for any reason within 30 days following placement.
Incidence of PICC-related complications before day 30 | Up to day 30
  Incidence of PICC-related complications (infection, thrombotic event, obstruction, displacement requiring PICC replacement or not) in the 30 days following placement.

OTHER OUTCOMES:
Cost analysis in healthcare institutions | Up to day 30
  Costs related to consumption of care in healthcare institutions (hospitalisations for insertion and removal of PICC catheters, for complications related to PICC, etc.).
Cost analysis in the community | Up to day 30
  Identification of costs in the community on the basis of patient diaries.
Deterministic Sensitivity Analysis | Up to day 30
  Sensitivity analysis on main cost parameters represented graphically by tornado diagrams to analyze the impact of variations in key cost parameters.
Probabilistic Sensitivity Analysis | Up to day 30
  Sensitivity analysis represented by a 95% confidence interval to assess the robustness of the cost-effectiveness results.
Organisational impacts | Up to day 30
  Assessment of organisational impacts using a modelling tool to break down patient flows and a simulation tool to simulate scenarios in order to assess organisational needs and constraints.
Success rate of PICC placement strategy | Up to day 30
  Proportion of patients for whom PICC insertion was successful without major complications, as performance indicator
Total duration of medical interventions | Up to day 30
  Total time spent on medical interventions throughout the patient's care pathway, including initial application, re-dressing and management of complications, as performance indicator
Assessment of cost of care | Up to day 30
  Total costs of patient care, including hospital and community costs, as performance indicator

CONTACTS AND LOCATIONS:
Overall Officials: Grégoire WALLON, MD, Principal Investigator — Centre Leon Berard
Locations (1):
- Centre Léon Bérard, Lyon, France